CLINICAL TRIAL: NCT06111950
Title: Study of the Consequences of Mutations of the RNU4ATAC and RTTN Genes by Transcriptomic, Biochemical and Cellular Approaches in Order to Determine the Pathophysiology of Their Associated Syndromes: Microcephalic Osteodysplastic Primordial Dwarfism Type I/III, Roifman Syndrome and Lowry-Wood Syndrome
Brief Title: Study of the Pathophysiology of RNU4ATAC and RTTN Associated Syndromes
Acronym: ATAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL20_0599
Record Dates: First submitted 2023-03-31; First posted 2023-11-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Taybi Linder Syndrome; Microcephalic Osteodysplastic Primordial Dwarfism Types I and III; Roifman Syndrome; Lowry Wood Syndrome
Keywords: Genetic diseases; Splicing; Minor introns; U4atac; Primary cillium
MeSH Terms: conditions — Microcephalic osteodysplastic primordial dwarfism, type 1; Roifman syndrome; Lowry Wood syndrome; Genetic Diseases, Inborn | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RNU4ATAC patient (Other): Patient with bi-allelic mutation of the RNU4ATAC gene
  Interventions: Other: Blood samples; Other: Skin biopsies
- RNU4ATAC fetus (Other): Fetus with bi-allelic mutation of the RNU4ATAC gene
  Interventions: Other: Fetal samples
- RNU4ATAC parent (Other): Parent of patient or fetus with bi-allelic mutation of the RNU4ATAC gene and who present themselve mono-allelic mutation of the RNU4ATAC gene
  Interventions: Other: Blood samples
- RTTN patient (Other): Patient with bi-allelic mutation of the RTTN gene
  Interventions: Other: Blood samples; Other: Skin biopsies
- RTTN fetus (Other): Fetus with bi-allelic mutation of the RTTN gene
  Interventions: Other: Fetal samples

INTERVENTIONS:
Other: Blood samples — Blood samples of 5 ml to 15 ml depending on their weight
  Arms: RNU4ATAC parent; RNU4ATAC patient; RTTN patient
Other: Skin biopsies — Biopsies of fragment of skin 2 to 3 mm long by 1 mm wide and 1 mm deep will preferably be taken on the inside of the arm, in the upper third, between the bend of the elbow and the hollow of the armpit under strict sterility conditions.
  Arms: RNU4ATAC patient; RTTN patient
Other: Fetal samples — Skin, muscle, brain and bone biopsies will be collected from fetuses in the autopsy room after the medical termination of pregnancy or miscarriage
  Arms: RNU4ATAC fetus; RTTN fetus

SUMMARY:
In the human genome, about 750 genes contain one intron excised by the minor spliceosome. These genes are named U12 genes, and these introns, minor or U12 introns. The minor spliceosome comprises its own set of snRNAs, among which U4atac. Its non-coding gene, RNU4ATAC, has been found mutated in Taybi-Linder (TALS), Roifman (RFMN) and Lowry-Wood syndromes (LWS). These rare developmental disorders associate ante- and post-natal growth retardation, microcephaly, skeletal dysplasia, intellectual disability, retinal dystrophy and immunodeficiency. Their physiopathological mechanisms remain unsolved: the number of U12 genes involved, their identity and function, or the cellular mechanisms impacted by the splicing defect, are still unknown.

The hypothesis of the study is that U12 genes coding for primary cilia components are particularly sensitive to minor splicing defects caused by RNU4ATAC mutations. Indeed, a child showing signs of TALS but negative for RNU4ATAC was found to carry a homozygous variant in the RTTN gene, coding for the rotatin protein located at the centrosome and the base of the primary cilia and playing a role in maintaining these structures. In addition, bi-allelic RNU4ATAC mutations were identified in five patients presenting with traits suggestive of the Joubert syndrome (JBTS), a well-characterized ciliopathy. These patients also present with traits typical of TALS/RFMN/LWS.

To better understand the causes of these pathologies, a cohort of patients with syndromes associated with bi-allele mutations of the RNU4ATAC or RTTN gene will be gathered, in order to conduct studies on the cells of these patients. Blood samples will be taken, as well as skin biopsies, if possible. These samples will be used to create induced pluripotent stem cell lines. Blood samples will also be collected from the parents of RNU4ATAC patients, to eliminate in transcriptomic analyses expression variations due to differences in genetic background. Biopsies of skin, muscle and brain tissue will be collected on foetuses carrying two-allele RNU4ATAC or RTTN mutations whose parents have had a miscarriage or have chosen to have a medical abortion. The biological samples collected will be used to study the transcription level of U12 genes, the splicing of their pre-messenger RNA, their main cellular functions, and the structural characteristics of tissues and cells.

ELIGIBILITY:
Inclusion Criteria:

TALS, RFMN, LWS or other pathology patients

* Woman or man
* All ages
* Presence of bi-allelic mutations of RNU4ATAC or RTTN
* Written consent of parents or legal guardian(s)
* Affiliation to a Social Security scheme

Healthy participants (Parent of the patient)

* Woman or man
* Major
* Presence of mono-allelic mutations of RNU4ATAC
* Written consent of the participant
* Affiliation to a Social Security scheme

Parents having recourse to a medical termination of pregnancy or having had a spontaneous miscarriage (for fetus samples)

* Woman or man
* Major
* Presence of bi-allelic mutations of RNU4ATAC or RTTN in the fetus
* Written parental consent
* Affiliation to a Social Security scheme

Exclusion Criteria:

Subject participating in another research including an exclusion period still in progress.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2029-08-27 (Estimated); Study Completion 2029-08-27 (Estimated)

PRIMARY OUTCOMES:
Identification of RNU4ATAC mutations consequences at the cellular level | 5 years
  The dysfunctions present in the different cell types obtained from RNU4ATAC patients will be identified by comparison with the controls, and will be compared with those present in RTTN patients.
  Consequences in cells of patients of RNU4ATAC mutations on the length and the structure of the primary cilium, as measured by fluorescence microscopy, and on the formation of small nuclear ribonucleoprotein (snRNPs) particles, as measured by glycerol gradient sedimentation analysis

SECONDARY OUTCOMES:
Minor splicing anomalies | 5 years
  The number and list of U12 genes for which an alteration of splicing will be identified in patient cells relatively to control cells will be compared, taking into account the different phenotypes (TALS, RFMN, LWS and other pathologies possibly identified).
  Consequences in cells of patients of RNU4ATAC mutations on minor intron splicing, as measured by intron retention analysis with the IRFinder and KisSplice bioinformatics softwares following RNA-sequencing experiments
Understanding of neuronal differentiation anomalies | 5 years
  Abnormalities in the behaviour of cells differentiated into neuronal progenitors will be identified by comparison with the controls, and will be compared taking into account the different phenotypes (TALS, RFMN, LWS and other pathology(s)) possibly identified).
  Consequences of RNU4ATAC mutations on the ability of induced pluripotent stem cells to differentiate towards the neuronal lineage, as measured by immunocytochemistry

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre de référence des anomalies du développement et syndromes malformatifs du Sud-Ouest Occitanie Réunion, CHU de Bordeaux-GH Pellegrin, Bordeaux
  - Centre de référence anomalies du développement de Lyon, Hôpital Femme Mère Enfant, Bron
  - Centre de référence des anomalies du développement et syndromes malformatifs de l'Est, CHU de DIJON, Dijon
  - Centre de référence des anomalies du développement et syndromes malformatifs de l'inter région Nord-Ouest, Hôpital J de Flandre, Lille
  - Unité Fonctionelle d'embryo-fœtopathologie, Hôpital Necker-Enfants Malades, Paris
  - Centre de référence des anomalies du développement et syndromes malformatifs de l'Ouest, Hôpital Sud, Rennes

IPD SHARING:
Plan to Share IPD: No